CLINICAL TRIAL: NCT01597466
Title: A Comparison Study of Two Different Techniques for Identifying the Epidural Space in Patients Requiring Thoracic Epidural Analgesia: a Prospective Multicentric Randomized Study
Brief Title: Epidrum for Thoracic Epidural Analgesia
Acronym: Epidrum-Tho
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012/01; 2012-A00083-40 (Other: ANSM)
Record Dates: First submitted 2012-05-05; First posted 2012-05-14 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epidrum (Experimental): Epidrum (Exmoor Innovations, Lisieux Way, Taunton, Somerset TA1 2LB, U.K.)
  Interventions: Device: Epidural catheter placement
- Loss of resistance technique (Active Comparator)
  Interventions: Procedure: Epidural catheter placement

INTERVENTIONS:
Device: Epidural catheter placement — Epidural space is located using Epidrum (Exmoor Innovations, Lisieux Way, Taunton, Somerset TA1 2LB, U.K.)
  Arms: Epidrum
Procedure: Epidural catheter placement — Epidural space is located using loss of resistance technique (saline solution)
  Arms: Loss of resistance technique

SUMMARY:
The purpose of this study is to evaluate the use of the Epidrum device to identify the epidural space in patients requiring thoracic epidural analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Elective major thoracic surgery requiring thoracic epidural analgesia

Exclusion Criteria:

* Contraindication to epidural anesthesia
* Marked spinal deformities or a history of spinal instrumentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Ease to identify the epidural space | 30 minutes
  Number of cases having required more than 2 punctures and number of failures of the technique

SECONDARY OUTCOMES:
Duration of epidural procedure | 30 minutes
Number of cutaneous punctures | 30 minutes
Number of needle redirections | 30 minutes
Ease of epidural catheter insertion | 30 minutes
Number of inadequate postoperative analgesia | one day after anesthesia
  asymmetric, incomplete or failed analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Morgan Le Guen, MD, Principal Investigator — Hopital Foch; Marc Fischler, MD, Study Chair — Hopital Foch
Locations (2):
- France (2):
  - CHU Marseille, Marseille
  - Hopital Foch, Suresnes